# Microvascular Sex and Age-related Day-to-day Variability in Healthy Subjects

- Statistical Analysis plan

NCT-number: 06009939

### Document revision history

| Issue | Summary of change |
|-------|-------------------|
| 01 | New document |

#### Statistical program

The statistical analysis will be conducted in IBM SPSS (SPSS, Chicago, IL).

#### Statistical analysis of Day-to-day variability

Median values from the baseline data of each measurement will be extracted for all parameters. The maximum value during the post-occlusive reactive hyperemia (PORH) will also be extracted for all parameters. See Table 1 and Table 2 for more details regarding which values will be included in the data analysis.

Table 1. Values extracted from the EPOS data of each measurement.

| Time period | Conventiona<br>I perfusion | Speed-<br>resolved-<br>perfusion<br>-Low speed | Speed-<br>resolved-<br>perfusion<br>-Medium<br>speed | Speed-<br>resolved-<br>perfusion<br>-High speed | Oxygen<br>saturation | Vessel<br>diameter | RBC tissue<br>fraction |
|---|---|---|---|---|---|---|---|
| Baseline of foot (10 minutes) | Median | Median | Median | Median | Median | Median | Median |
| Occlusion of foot (5 minutes) | No value extracted | No value extracted | No value extracted | No value extracted | No value extracted | No value<br>extracted | No value extracted |
| PORH in foot<br>(5 minutes) | Peak value | Peak value | Peak value | Peak value | Peak value | Peak value | Peak value |
| Baseline of arm (10 minutes) | Median | Median | Median | Median | Median | Median | Median |
| Occlusion of arm (5 minutes) | No value extracted | No value extracted | No value extracted | No value extracted | No value extracted | No value<br>extracted | No value extracted |
| PORH in arm<br>(5 minutes) | Peak value | Peak value | Peak value | Peak value | Peak value | Peak value | Peak value |

Table 2. Values extracted from the PSI-X camera of each measurement.

| Time period | Conventional perfusion | Speed-resolved-<br>perfusion<br>-Low speed | Speed-resolved-<br>perfusion<br>-Medium speed | Speed-resolved-<br>perfusion<br>-High speed | Oxygen saturation |
|---|---|---|---|---|---|
| Baseline of foot (10 minutes) | Median | Median | Median | Median | Median |
| Occlusion of foot (5 minutes) | No value extracted | No value extracted | No value extracted | No value extracted | No value extracted |
| PORH in foot<br>(5 minutes) | Peak value | Peak value | Peak value | Peak value | Peak value |
| Baseline of arm (10 minutes) | Median | Median | Median | Median | Median |
| Occlusion of arm (5 minutes) | No value extracted | No value extracted | No value extracted | No value extracted | No value extracted |
| PORH in arm<br>(5 minutes) | Peak value | Peak value | Peak value | Peak value | Peak value |

To identify potential sex- and age-related variability, Wilcoxon test will be conducted for non-normally distributed data and t-test for normally distributed data. To compare the data collected from the foot to the arm, Kruskal-Wallis or Anova will be used.

Since multiple comparisons between groups will be conducted, Bonferroni corrections will be done to reduce the risk of Type 1 error.

#### Statistical analysis of Vasomotion data

Table 3 describes the values from each measurement which will be included in the flowmotion analysis. The columns describe the different flowmotion signal types, the rows describe the different groups which will be compared.

| Table 3. Values extracted for the flowmotion analysis, from each m | ch measurement. |
|---|---|
|---|---|

| | Cardiac | Respiratory | Myogenic | Neurogenic | Endothelial |
|---|---|---|---|---|---|
| Baseline of foot (10 minutes) | Mean-energy over time | Mean-energy over time | Mean-energy over time | Mean-energy over time | Mean-energy over time |
| Occlusion of foot (5 minutes) | Mean-energy over time | Mean-energy over time | Mean-energy over time | Mean-energy over time | Mean-energy over time |
| PORH in foot<br>(5 minutes) | Mean-energy over time | Mean-energy over time | Mean-energy over time | Mean-energy over time | Mean-energy over time |
| Baseline of arm (10 minutes) | Mean-energy over time | Mean-energy over time | Mean-energy over time | Mean-energy over time | Mean-energy over time |
| Occlusion of arm (5 minutes) | Mean-energy over time | Mean-energy over time | Mean-energy over time | Mean-energy over time | Mean-energy over time |
| PORH in arm (5 minutes) | Mean-energy over time | Mean-energy over time | Mean-energy over time | Mean-energy over time | Mean-energy over time |

Flowmotion analysis is described in depth in the following articles:

- Fredriksson et al. 2021, Vasomotion analysis of speed resolved perfusion, oxygen saturation, red blood cell tissue fraction, and vessel diameter: Novel microvascular perspectives.
- Hultman et al. 2023, Flowmotion imaging analysis of spatiotemporal variations in skin microcirculatory perfusion.

Please see references for further details.

For the time being, the different flowmotion signals will be compared on a group level.

#### Significance level

Significance level is set to p < 0.05.

#### Method for dealing with missing data

The goal is to have 48 complete set of data collection for the variability analysis and recruitment to the study will continue until this is achieved. Flowmotion analysis is more sensitive to artefacts, which most likely will be discovered late in the process once the recruitment to the study already is complete. Therefore we expect to exclude some measurements and most likely will not reach 48 complete sets of flowmotion signals.

#### Motivation to the number of study-participants

12 participants in each group (men and women, age 20-30 years or 50-60 years), which adds up to a total of 48 participants, is chosen due to the tradition within the study field. In addition, we do not know if there is a difference among the four groups, which is why we chose a smaller study population.

#### Method for dealing with outliers

Outliers in the collected data caused by movement (and thereby considered artifacts) will be handled using the algorithm presented in reference 2 above.

## Visual presentation of data

Data as well as our findings will be presented with boxplots or regression plots.